CLINICAL TRIAL: NCT01201252
Title: An Observational, Hospital-based Surveillance to Estimate the Disease Burden of Acute Rotavirus (RV) Gastroenteritis (GE) in Children < 5 Years of Age in United Arab Emirates (UAE).
Brief Title: Study to Estimate the Disease Burden of Acute Rotavirus Gastroenteritis in Children < 5 Years in United Arab Emirates
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 110846
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Rotaviral Gastroenteritis
Keywords: children; gastroenteritis; Rotavirus
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool

GROUPS / COHORTS (1):
- Acute gastroenteritis Group: Suspected/confirmed cases of rotavirus gastroenteritis in children < 5 years of age
  Interventions: Procedure: Stool sampling

INTERVENTIONS:
Procedure: Stool sampling — Stool samples will be collected, tested and genotyped for the presence of rotavirus

SUMMARY:
The purpose of this study is to estimate the disease burden and epidemiology of rotavirus gastroenteritis in children less than 5 years of age, in United Arab Emirates. Acute gastroenteritis cases will be identified from acute gastroenteritis hospitalisation log book and stool samples will be collected from all suspected and confirmed acute gastroenteritis cases.

ELIGIBILITY:
Inclusion Criteria:

* A male or female < 5 years of age at the time of admission to the study hospital for acute gastroenteritis.
* Written informed consent obtained from the parent or guardian of the subject.

Exclusion Criteria:

* The diagnosis for treatment at the study site does not include acute gastroenteritis.
* The onset of acute gastroenteritis after admission to the hospital i.e. 48 hours after hospital admission.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children < 5 years of age hospitalised with acute gastroenteritis
Sampling Method: Non-Probability Sample
Enrollment: 717 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of diarrhoeal hospitalisations in children < 5 years of age, which are attributable to rotavirus. | Twelve months from study initiation

SECONDARY OUTCOMES:
Age and seasonal distribution of hospitalisations associated with rotavirus in children < 5 years of age. | Twelve months from study initiation
Occurrence of intravenous re-hydration treatment and/or other treatments due to rotavirus gastroenteritis. | Twelve months from study initiation
Distribution of different strains of rotavirus in children < 5 years of age. | Twelve months from study initiation
Occurrence of acute gastroenteritis and rotavirus gastroenteritis among all hospitalisations of children < 5 years of age. | Twelve months from study initiation
Occurrence of severe dehydrating rotavirus gastroenteritis based on Vesikari scale among children < 5 years of age. | Twelve months from study initiation

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United Arab Emirates (3):
  - GSK Investigational Site, Abu Dhabi
  - GSK Investigational Site, Al Ain City
  - GSK Investigational Site, Sharjah city